CLINICAL TRIAL: NCT01209689
Title: A Randomized, Double-blind, Parallel Group Placebo-controlled Study of the Safety and Reduction of Signs and Symptoms During Treatment With Tocilizumab (TCZ) Versus Placebo in Patients With Ankylosing Spondylitis Who Have Had an Inadequate Response to Previous TNF Antagonist Therapy
Brief Title: A Study of Tocilizumab (RoActemra/Actemra) in Patients With Ankylosing Spondylitis Who Have Had an Inadequate Response to Previous Tumor Necrosis Factor (TNF) Antagonist Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Clinical development program terminated due to failure to achieve efficacy
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA22908; 2009-017488-40
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2012-12

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Tocilizumab 4 mg/kg (Experimental): Patients received tocilizumab 4 mg/kg intravenously every 4 weeks for 24 weeks.
  Interventions: Drug: Tocilizumab
- Tocilizumab 8 mg/kg (Experimental): Patients received tocilizumab 8 mg/kg intravenously every 4 weeks for 24 weeks.
  Interventions: Drug: Tocilizumab
- Placebo (Placebo Comparator): Patients received placebo to tocilizumab intravenously every 4 weeks for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab
  Other Names: RoActemra; Actemra
  Arms: Tocilizumab 4 mg/kg; Tocilizumab 8 mg/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled study evaluated the safety and efficacy of tocilizumab (RoActemra/Actemra) in patients with ankylosing spondylitis (AS) who had an inadequate response to previous tumor necrosis factor (TNF) antagonist therapy. Patients were randomized to receive tocilizumab at a dose of either 8 mg/kg or 4 mg/kg intravenously (iv) or placebo every 4 weeks for 24 weeks. The double-blind treatment period was followed by open-label treatment with tocilizumab 8 mg/kg iv every 4 weeks until Week 104 for all patients.

This study and all further clinical development of tocilizumab AS was halted after a review of 12-week data from Study NA22823, a randomized double-blind, placebo-controlled study in TNF antagonist naïve AS patients, failed to demonstrate efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age.
* Ankylosing spondylitis as defined by the modified New York criteria for ≥ 3 months prior to baseline.
* Active disease at screening and baseline (Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] ≥ 4.0, spinal pain visual analog scale [VAS] ≥ 40).
* Inadequate response or intolerant to 1 or more previous non-steroidal anti-inflammatory drugs (NSAIDs).
* Inadequate response to treatment with etanercept, infliximab, adalimumab, or golimumab because of inadequate efficacy.
* Tumor necrosis factor (TNF) antagonist therapy must have been discontinued at least 8 weeks prior to baseline (etanercept 4 weeks).
* Traditional disease-modifying anti-rheumatic drugs (DMARDs) must be withdrawn for at least 4 weeks prior to baseline (methotrexate, sulfasalazine, and hydroxychloroquine or chloroquine may be allowed if at stable dose for at least 4 weeks prior to baseline).
* Oral corticosteroids (≥ 10 mg/day prednisone or equivalent) and NSAIDs/cyclooxygenase-2 [COX-2] inhibitors must be at stable dose for at least 4 weeks prior to baseline.

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months after randomization.
* Total ankylosis of spine (as determined by investigator).
* Inflammatory rheumatic disease other than ankylosing spondylitis.
* Active, acute uveitis at baseline.
* Previous treatment with tocilizumab.
* Intra-articular or tendon injections or parenteral corticosteroids within 4 weeks prior to screening.
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
* Active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infection.
* History of or currently active primary or secondary immunodeficiency.
* Body weight > 150 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (125):
- United States (19):
  - Huntington Beach, California
  - Aventura, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Idaho Falls, Idaho
  - Wichita, Kansas
  - Hagerstown, Maryland
  - Saint Claire Shores, Michigan
  - Freehold, New Jersey
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Duncansville, Pennsylvania
  - Austin, Texas
  - Houston, Texas
- Australia (4):
  - Heidelberg
  - Hobart
  - Sydney
  - Woodville
- Belgium (5):
  - Brussels
  - Ghent
  - Kortrijk
  - Liège
  - Yvoir
- Brazil (3):
  - Cuiabá
  - Goiânia
  - São Paulo
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Canada (10):
  - Calgary, Alberta
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Mississauga, Ontario
  - St. Catharines, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Trois-Rivières, Quebec
  - St. John's
- Czechia (6):
  - Bruntál
  - Hlučín
  - Olomouc
  - Prague
  - Uherské Hradiště
  - Zlín
- Denmark (3):
  - Esbjerg
  - Hellerup
  - Vejle
- France (13):
  - Besançon
  - Bordeaux
  - Boulogne-Billancourt
  - Créteil
  - Grenoble
  - Le Kremlin-Bicêtre
  - Lyon
  - Montpellier
  - Orléans
  - Paris
  - Rouen
  - Strasbourg
  - Vandœuvre-lès-Nancy
- Germany (14):
  - Berlin
  - Cologne
  - Erlangen
  - Frankfurt
  - Gommern
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - München
  - Regensburg
  - Rostock
  - Tübingen
  - Würzburg
- India (4):
  - Bangalore
  - Jaipur
  - New Delhi
  - Secunderabad
- Italy (9):
  - Ferrara
  - Florence
  - Monserrato
  - Padua
  - Pisa
  - Prato
  - Reggio Emilia
  - Roma
  - Siena
- Lithuania (2):
  - Kaunas
  - Klaipėda
- Amsterdam, Netherlands
- Poland (7):
  - Bydgoszcz
  - Krakow
  - Lublin
  - Poznan
  - Torun
  - Warsaw
  - Wroclaw
- Slovakia (2):
  - Košice
  - Piešťany
- South Africa (5):
  - Cape Town
  - Durban
  - Pinelands
  - Pretoria
  - Stellenbosch
- Spain (8):
  - A Coruña
  - Alcorcón
  - Barcelona
  - Córdoba
  - Lugo
  - Madrid
  - Oviedo
  - Sabadell
- United Kingdom (8):
  - Basingstoke
  - Bath
  - Greenock
  - Leeds
  - London
  - Salford
  - Stoke-on-Trent
  - Wigan

REFERENCES:
- [Derived] Sieper J, Porter-Brown B, Thompson L, Harari O, Dougados M. Assessment of short-term symptomatic efficacy of tocilizumab in ankylosing spondylitis: results of randomised, placebo-controlled trials. Ann Rheum Dis. 2014 Jan;73(1):95-100. doi: 10.1136/annrheumdis-2013-203559. Epub 2013 Jun 13. PMID 23765873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Because of the early termination of the study and the limited and varying duration of treatment, the 4 mg/kg and 8 mg/kg tocilizumab dose groups were combined in the efficacy and safety analyses and reporting.
Groups:
- Tocilizumab 4 or 8 mg/kg: Patients received tocilizumab 4 or 8 mg/kg intravenously every 4 weeks for 24 weeks.
Period: Overall Study
Arm/Group | Tocilizumab 4 or 8 mg/kg | Placebo
Started | 91 | 22
Completed | 0 | 0
Not Completed | 91 | 22
Not completed — Insufficient Therapeutic Response | 7 | 2
Not completed — Refused Treatment | 8 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Violation of Selection Criteria at Entry | 1 | 0
Not completed — Failure to Return | 3 | 0
Not completed — Sponsor's Decision to Stop the Study | 68 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab 4 or 8 mg/kg | Placebo | Total
Number analyzed (Participants) | 91 | 22 | 113
Age Continuous [Mean (Standard Deviation); unit: years] | 44.1 (12.08) | 45.0 (12.66) | 44.3 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 8 | 37
  Male | 62 | 14 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of ASsessment in Ankylosing Spondylitis 20 (ASAS20) Responders at Week 12
Description: ASAS20 was defined as an improvement of ≥ 20% and an absolute improvement of ≥ 10 units on a 0-100 visual analog scale (VAS) from Baseline to Week 12 in 3 of 4 domains: 1-Patient global assessment (with extremes labelled none and severe), 2-Pain assessment (average total and nocturnal pain scores with extremes labelled no pain and most severe pain), 3-Function (represented by the Bath Ankylosing Spondylitis (BAS) Functional Index [BASFI] average of 10 questions regarding ability to perform specific tasks with extremes labelled easy and impossible), and 4-Inflammation (average of the last 2 questions on the 6-question BAS Disease Activity Index [BASDAI] concerning morning stiffness intensity with extremes labelled none and very severe and duration between 0 and 2 or more hours); and the absence of deterioration (of at least 20% and absolute change of at least 10 units on a 0-100 mm scale) in the remaining domain.
Time Frame: Baseline to Week 12
Population: Intent-to-treat population: All randomized patients who received at least 1 dose of treatment. The analysis only included assessments while patients were receiving double-blind treatment and that occurred prior to withdrawal or the date when all patients were unblinded (15 Jul 2011). Patients who withdrew or escaped were considered non-responders.
Measure: Number; unit: Percentage of patients
Arm/Group | Tocilizumab 4 or 8 mg/kg | Placebo
Number analyzed (Participants) | 79 | 21
Percentage of patients | 12.7 | 14.3

ADVERSE EVENTS:
Time Frame: For the tocilizumab group, adverse events (AE) were reported from randomization to the end of the study. For the placebo group, AEs were reported from randomization only until participants escaped or switched to tocilizumab.
Description: Safety population: Patients who received at least 1 dose of study medication and had at least 1 post-baseline safety assessment. Patients were assigned to groups as treated; 95 patients in the combined tocilizumab groups, including 4 patients randomized to placebo who received escape therapy of 8 mg/kg tocilizumab at Week 16.
Groups:
- Tocilizumab: Patients randomized to tocilizumab who received intravenous infusions of 4 mg/kg or 8 mg/kg tocilizumab once every 4 weeks for 24 weeks and patients randomized to placebo who switched or escaped to tocilizumab treatment.
Arm/Group | Tocilizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 6/95 | 0/22
Other Adverse Events (participants affected / at risk) | 6/95 | 1/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=95) | Placebo (N=22)
Anaphylactic reaction (Immune system disorders) | 2 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pasteurella infection (Infections and infestations) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=95) | Placebo (N=22)
Headache (Nervous system disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.